CLINICAL TRIAL: NCT06800976
Title: Study of Cognitive and Behavioural Biases in People With Idiopathic Environmental Intolerance (IEI) Versus Healthy Controls
Acronym: BELIEFS VS
Status: Not yet recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C24-26
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers; Idiopathic Environmental Intolerance
Keywords: predictive processing; Mechanisms; symptoms associated with environmental factors; negative affect
MeSH Terms: conditions — Multiple Chemical Sensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy: Healthy participants with no idiopathic environmental intolerance

SUMMARY:
Symptoms that patients attribute to the environment when no environmental cause can be identified are known as "idiopathic environmental intolerance" (IEI). IEI is often associated with a major psychological and socio-professional impact. Specific diagnostic tools and evidence-based treatment programs are still lacking. As a result, IEI patients often feel left behind by physicians and public health policies.

A number of environmental agents are singled out by IEI sufferers, including chemicals (cleaning products, tobacco smoke), electromagnetic fields generated by cell phones and base stations, air conditioning and infrasound emitted by wind turbines. Patients hold one or more of these environmental agents responsible for a very wide range of chronic, non-specific physical symptoms such as diffuse pain, fatigue, dizziness, dyspnoea, hot flushes, nausea, tinnitus or palpitations, but also cognitive symptoms such as loss of memory or concentration. However, the medical examination of IEI patients shows no evidence of bodily dysfunction.

Furthermore, numerous exposure studies have shown that environmental agents did not alter the biological parameters of IEI patients, that patients could not reliably distinguish between real and fictitious exposures, and that they only presented symptoms when they thought the exposure was real, whether this was true or not. This suggests that IEI symptoms can be considered "functional", resulting from an alteration in the way the body is felt rather than from injury to the body itself. Recently, several authors including Lemogne and Pitron have proposed a cognitive model of body awareness and more specifically of functional physical symptoms.This model is part of a Bayesian understanding of brain function, which is increasingly seen as a process underlying all perceptual experiences.From this perspective, bodily experiences are the result of probabilistic calculations Two sources of information are integrated, weighted by their reliability (accuracy) with regard to the current context: the body's sensory signals on the one hand (i.e. peripheral nerve inputs) and "priors" about the body on the other (i.e. pre-existing information from previous bodily experiences, beliefs about the body, emotions, etc.). In functional physical symptoms, it has been suggested that priors override the body's sensory signals, thus skewing bodily perception.This would be the consequence of an imbalance between low-precision sensory signals on the one hand, and high-precision priors on the other.

In line with this model, Van den Bergh and Witthöft have proposed an understanding of IEI as arising from a nocebo effect.Here, we propose a research project with patients suffering from IEI to test and validate this Bayesian theoretical model of IEI, the main study C22-19, BELIEFS which is currently recruiting.

This ancillary study, C24-26 BELIEFS-VS, enables us to include a population of healthy volunteers whom we will compare with the IEI patients in the main C22-19 BELIEFS study.

DETAILED DESCRIPTION:
In the main BELIEFS study (ClinicalTrials ID NCT05973214), we are investigating the efficacy of a dedicated CBT treatment program for people with IEI, and the evolution of cognitive biases before versus after the treatment program. The present BELIEFS-VS ancillary study aims to include a group of healthy volunteers in order to compare cognitive outcomes in people with IEI. This BELIEFS-VS ancillary study will enable us to better study the cognitive characteristics of IEI patients in comparison with non-affected individuals, and thus gain a better understanding of the pathophysiology of the condition.

Methods and Analysis:

This is an observational study. Healthy controls will be age- and gender-matched to IEI patients. The healthy controls will be invited to one in-person session in our facilities, where they will be asked to fill in some questionnaires and complete some tasks (the Affective Picture Paradigm and the Belief Updating Task).

Ethics and dissemination:

Ethics approval has been granted. Results from this study will be published in peer-reviewed journals and presented at international conferences.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older; not suffering from an idiopathic environmental intolerance; informed consent is given.

Exclusion Criteria:

* Suffering from a current psychiatric or neurological condition
* not being fluent in spoken and written French
* person subject to a period of exclusion for other research
* being imprisoned/jailed
* being hospitalized
* Persons of legal age who are subject to a legal protection measure (e.g. conservatorship, guardianship), persons of legal age who are unable to express their consent and who are not subject to a protection measure.
* being pregnant or breast-feeding

Translated with DeepL.com (free version)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We are recruiting healthy participants that will be age- and gender-matched to participants in the BELIEFS study, who live with idiopathic environmental intolerances.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Performance on the Belief Updating Task | (Single assessment)
Performance on the Affective Picture Paradigm | (Single assessment)

SECONDARY OUTCOMES:
The Somatic Symptom Disorder - B Criteria Scale | (Single Assessment)
  Measures the B criterion for Somatic Symptom Disorder (SSD) and symptom burden: The total score ranges between 0 and 48, with a higher score reflecting higher levels of the psychological features of the SSD, or worse outcome.
Symptom Interpretation Questionnaire | (Single Assessment)
  Measures causal attributions individuals make of common somatic symptoms by using three sub scales: somatic (range 13-36), psychological (range: 13-52), and environmental/normalizing (range: 17-49). Each sub score represents the extent with which each sub scale is endorsed as a possible cause for symptoms (higher score means higher outcome).
Modern Health Worries Scale short (12-item) version | (Single Assessment)
  Measures Modern Health Worries (concerns of respondents about modern environmental issues/threats of modernity). Scores range from 12 to 60 with higher scores indicating more concern or worse outcome.
Climate Change Anxiety Scale | (Single Assessment)
  Measures Climate Change Anxiety with scores ranging from 13 to 65 and higher scores indicating higher levels of climate change anxiety, or worse outcome.
Hospital Anxiety and Depression scale | (Single Assessment)
  Measures Depression and Anxiety. Score ranges from 0 to 21 per subscale with higher score representing worse outcome.
Short Form Health Survey - 12 | (Single Assessment)
  Measures quality of life with a minimum value of zero and a maximum value of 100. Higher score indicates better outcome.
Body Perception Questionnaire - Very Short Form | (Single Assessment)
  Measures body awareness and autonomic stress response patterns. Scores range from 12 to 60. Particularly high scores may indicate the autonomic nervous system is frequently activated by stress or chronic threat responses (i.e. worse outcome)
Levels of Emotional Awareness Scale 10 item | (Single Assessment)
  Measures the Level of Emotional Awareness with a maximum score of 50. Higher scores indicating greater awareness and differentiation in emotions, or better outcome.
Short version of the Intolerance of Uncertainty Scale | (Single Assessment)
  Measures Intolerance to Uncertainty with total scores ranging from 12 to 60 with higher score representing worse outcome. The total scores encompasses two sub-scales: prospective anxiety and inhibitory anxiety. A greater score in each subscale indicates a greater level of prospective anxiety and inhibitory anxiety.
Number and intensity of physical symptoms - QEESI (subsection symptoms) | (Single Assessment)
  This subscales measures various physical symptoms one might experience in everyday life. Participants can score between 0 and 100 points, with a higher score indication more and more intense symptoms (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Cédric Lemogne, Dr., Principal Investigator — APHP Hôtel-Dieu
Locations (1):
- Unité de pathologies professionnelles et environnementales, Hôtel-Dieu, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided